CLINICAL TRIAL: NCT01837667
Title: A Phase I Study of Intravenous LB-100 for Injection as a Single Agent and in Combination With Docetaxel in the Treatment of Patients With Advanced Solid Tumors
Brief Title: Phase I Study of LB-100 With Docetaxel in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lixte Biotechnology Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L12-20661
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-09

CONDITIONS: Tumors; Neoplasms; Cancer
MeSH Terms: conditions — Neoplasms | interventions — LB100; Injections; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LB-100 for Injection and Docetaxel (Experimental): Part 1: LB-100 infusion. Part 2: LB-100 infusion and docetaxel infusion.
  Interventions: Drug: LB-100 for Injection; Drug: Docetaxel

INTERVENTIONS:
Drug: LB-100 for Injection — Part 1 and Part 2: LB-100 for Injection infusion on Days 1,2,3 of each 21 day cycle.
Drug: Docetaxel — Part 2: Docetaxel infusion on Day 2 of each 21 day cycle.
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to test the safety of an investigational drug called LB-100 for Injection for treatment of solid tumors, when given with or without docetaxel. LB-100 is a small molecule that in laboratory and animal studies has shown activity when used by itself or together with drugs approved to treat some types of cancer (chemotherapeutic agents). Docetaxel is a drug that has been approved for the treatment of some types of cancer; one of the trade names for docetaxel is Taxotere®. The study is in 2 parts. Part 1: Patients will receive injections of LB-100. Part 2: Patients will receive injections of LB-100 and docetaxel. This is the first study where LB-100 for Injection will be used in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Part 1 only: Patients with histologically or cytologically proven progressive or metastatic solid tumors who have failed standard treatment and have no other effective treatment available.

   Part 2 only: Patients with histologically or cytologically proven progressive or metastatic solid tumors who have failed standard treatment and have no other effective treatment available, or docetaxel-naive patients who have failed standard treatment and have tumors for which a docetaxel-based regimen would be appropriate.
2. Part 2 only: Patients must be docetaxel-naive.
3. Patients must have a life expectancy of at least 12 weeks.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Patients must be men and women >= 18 years of age.
6. Patients must have recovered from all acute adverse effects (excluding alopecia) of prior therapies to baseline or <= grade 1 prior to study entry.
7. Patients must have adequate bone marrow function, defined as an absolute neutrophil count >= 1.5 x 10^9/L and a platelet count >= 100 x 10^9/L.
8. Patients must have adequate renal function, defined as serum creatinine <= 1.5 x upper limit of normal (ULN) for the institution or a calculated creatinine clearance [Cockcroft-Gault method] must be >= 60 mL/min/1.73 m^2).
9. Patients must have adequate hepatic function, defined as:

   * Part 1 only: plasma total bilirubin <= 1.5 mg/dL, alanine transaminase (ALT) and aspartate transaminase (AST) <= 2.5 X ULN.
   * Part 2 only: plasma total bilirubin <= ULN; ALT and/or AST <= 1.5 X ULN concomitant with alkaline phosphatase <= 2.5 X ULN.
10. Female patients of childbearing potential must have a negative serum or urine pregnancy test result at time of pre-treatment screening.
11. Patients with reproductive potential must agree to use at least one form of barrier contraception prior to study entry and for up to 30 days beyond the last administration of study drug.
12. Patients must be capable of providing informed consent and must be willing to provide written informed consent prior to the start of any study-specific procedures.

Exclusion Criteria:

1. Patients may not have had prior chemotherapy, radiotherapy, hormonal therapy, or biologic therapy in the 4 weeks prior to study entry with the exception of mitomycin C or nitrosoureas, for which patients must be 6 weeks from prior treatment. For patients who have been treated with targeted therapy, 5 half-lives of that therapy (or 28 days, whichever is shorter) must have passed prior to enrollment in the study.
2. Part 2 only: Patients may not have had prior treatment with docetaxel.
3. Part 2 only: Patients with plasma total bilirubin > ULN; ALT and/or AST > 1.5 X ULN concomitant with alkaline phosphatase > 2.5 X ULN.
4. Patients may not have any concomitant condition that could compromise the objectives of this study and the patients' compliance and ability to tolerate this therapy and complete at least 2 cycles of therapy, including, but not limited to the following:

   * Congestive heart failure or uncontrolled angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension, or dysrhythmias.
   * Active infection.
   * Unstable diabetes mellitus.
   * Psychiatric disorder that may interfere with consent and/or protocol compliance.
   * Uncontrolled seizure activity.
   * Prior history of inflammatory bowel disease.
   * Prior history of pulmonary fibrosis.
   * Prior history of cardiomyopathy.
5. Patients with a history of central nervous system (CNS) malignancy.
6. Pregnant or breastfeeding women.
7. Patients with another malignancy in the past 3 years except: curatively treated non-melanoma skin cancer, or carcinoma in situ (either cervix or breast) that does not require further treatment.
8. Patients with known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
9. Part 2 only: Patients with a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80 (for example, drugs formulated with polysorbate 80 include, but are not limited to: Aranesp, Eprex, Cordarone, some vaccines).
10. Part 2 only: Patients with >= grade 2 peripheral neuropathy.
11. Patients with an underlying diagnosis or disease state associated with an increased risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability of LB-100 for Injection treatment plus docetaxel. | Starting from date of first dose up to 30 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, MD, FACP, Principal Investigator — City of Hope National Medical Center; Aaron Mansfield, MD, Principal Investigator — Mayo Clinic; Fadi Braiteh, MD, Principal Investigator — Comprehensive Cancer Centers of Nevada; Carlos Becerra, MD, Principal Investigator — Texas Oncology - Baylor Charles A Sammons Cancer Center; Donald Richards, MD, Principal Investigator — Texas Oncology - Tyler
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Tyler, Tyler, Texas

REFERENCES:
- [Result] Chung V, Mansfield AS, Braiteh F, Richards D, Durivage H, Ungerleider RS, Johnson F, Kovach JS. Safety, Tolerability, and Preliminary Activity of LB-100, an Inhibitor of Protein Phosphatase 2A, in Patients with Relapsed Solid Tumors: An Open-Label, Dose Escalation, First-in-Human, Phase I Trial. Clin Cancer Res. 2017 Jul 1;23(13):3277-3284. doi: 10.1158/1078-0432.CCR-16-2299. Epub 2016 Dec 30. PMID 28039265